CLINICAL TRIAL: NCT02328924
Title: There is a Cut Off Value of Luteinizing Hormone Predictive of in Vitro Fertilization Treatment Outcome? A Randomized Controlled Trial in Fixed Versus Flexible Gonadotropin-releasing Hormone Antagonist Protocols.
Brief Title: There is a Value of Luteinizing Hormone Predictive of in Vitro Fertilization Treatment Outcome in Antagonist Protocols?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: U.O.S. Procreazione Medicalmente Assistita e Congelamento Gameti (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Uospmacg
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LH value in fixed group (Other): LH value predictive of IVF in 104 patients entered in fixed protocol
  Interventions: Other: LH value
- LH value in flexible group (Other): LH value predictive of IVF in 109 patients entered in flexible protocols
  Interventions: Other: LH value

INTERVENTIONS:
Other: LH value — analyzed LH value in the the arms of the study, fixed and flexible protocols

SUMMARY:
This study, prospective randomized controlled trial, tried to identify a cut off value of luteinizing hormone predictive of in vitro fertilization outcome in a fixed or flexible gonadotropin-releasing hormone antagonist protocols.

202 norma-ovulatory women < 39 years were randomized to fixed or flexible group in GnRH antagonist protocols The follicular phase profile of luteinizing hormone, estradiol and progesterone in the two study groups was measured. Total number of retrieved oocytes, implantation and pregnancy rate were recorded.

.

ELIGIBILITY:
Inclusion Criteria:

* 1) age <39 years; (2) normal menstrual cycle (range of 26-32 days); (3) baseline follicle stimulating hormone levels < 12 IU/ml; (4) body mass index (BMI) between 18-30 Kg/m2; (5) no oral contraceptive pills taken in the last year

Exclusion Criteria:

* polycystic ovaries, age >39 years

Ages: 35 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
number of mature oocytes recruited after IVF with antagonist protocol | partecipant will be followed for the duration of the cycle of IVF and for the following three months